CLINICAL TRIAL: NCT06562582
Title: STunning in Acute Myocardial Infarction - Beta Blockers, Angiotensin Converting Enzyme Inhibitors and Sodium/Glucose Cotransporter 2 Inhibitors Trial A Low Intervention Clinical Tria
Brief Title: STunning in Acute Myocardial Infarction - BAS
Acronym: STAMI-BAS
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Vastra Gotaland Region (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: 2024-511789-35-00
Record Dates: First submitted 2024-08-16; First posted 2024-08-20 (Actual); Last update posted 2025-06-27 (Actual); Status verified 2024-08

CONDITIONS: Myocardial Infarct
Keywords: ST infarction; PCI; Bisoprolol; Ramipril; Dapagliflozin; Global longitudinal strain (GLS, %)
MeSH Terms: conditions — Myocardial Infarction | interventions — Bisoprolol; Angiotensin-Converting Enzyme Inhibitors; Sodium-Glucose Transporter 2 Inhibitors

STUDY DESIGN:
Intervention Model Description: This prospective, 2x2x2 factorial, randomized, controlled,
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (6):
- Bisoprolol (Active Comparator): Bisoprolol within 24 hours of PCI
  Interventions: Drug: Bisoprolol Oral Tablet
- No Bisoprolol (No Intervention): no beta blocker until day 7±12 hours
- Ramipril (Active Comparator): Ramipril within 24 hours of PCI
  Interventions: Drug: Ramipril Oral Product
- No Ramipril (No Intervention): no ramipril until day 7±12 hours after PCI
- Dapagliflozin (Active Comparator): Dapagliflozin within 24 hours versus
  Interventions: Drug: Dapagliflozin Oral Product
- No Dapagliflozin (No Intervention): no dapagliflozin treatment until day 7±12 hours after PCI

INTERVENTIONS:
Drug: Bisoprolol Oral Tablet — Timing of drug intervention after PCI
  Other Names: Betablocker
  Arms: Bisoprolol
Drug: Ramipril Oral Product — Timing of drug intervention after PCI
  Other Names: ACE inhibitor
  Arms: Ramipril
Drug: Dapagliflozin Oral Product — Timing of drug intervention after PCI
  Other Names: SGLT2 inhibitor
  Arms: Dapagliflozin

SUMMARY:
The objective of this trial is to examine the effect of immediate versus late administration of beta blockers, angiotensin converting enzyme inhibitors (ACEI), and sodium/glucose cotransporter 2 (SGLT2) inhibitors on echocardiographic parameters and biomarkers in subjects with ST-elevation myocardial infarction (STEMI)

DETAILED DESCRIPTION:
Left ventricular (LV) remodeling after ST-elevation myocardial infarction (STEMI) is associated with poor outcomes, but the mechanisms underlying adverse LV remodeling are poorly understood. It is also poorly understood how current guideline-recommended treatments affect early LV remodeling. This low interventional clinical trial will compare the effects of early versus late initiation of the three pharmacotherapies on early LV remodeling and cardiometabolic profiles.

Trial objective:

The objective of this trial is to examine the effect of immediate versus late administration of beta blockers, angiotensin converting enzyme inhibitors (ACEI), and sodium/glucose cotransporter 2 (SGLT2) inhibitors on echocardiographic parameters and biomarkers in subjects with ST-elevation myocardial infarction (STEMI).

Primary endpoint:

Global longitudinal strain (GLS, %) at day 7±24 hours after PCI, adjusted for baseline (day 0) GLS.

Trial design:

This prospective, 2x2x2 factorial, randomized, controlled, open-label, low intervention clinical trial will enroll subjects with STEMI who undergo primary percutaneous coronary intervention (PCI) within 6 hours of symptom onset.

Trial population:

Patients over the age of 18 with STEMI who undergo primary PCI

ELIGIBILITY:
Inclusion Criteria:

1. Patients with STEMI who undergo primary PCI within 6 hours of symptom onset (Excluding prodromal symptoms)
2. Informed consent

Exclusion Criteria:

1. Killip class ≥ 3
2. Chronic kidney disease with GFR < 25 ml/min/1.73 m2
3. Pre-existing non-reversible cardiac dysfunction or heart failure
4. Current treatment with any beta blocker, RAAS inhibitor or SGLT2 inhibitor
5. Absolute or relative contraindication to any one of the study drugs that confers a risk of patient safety if the patient participates in the trial and adheres to the protocol-specified recommendations, per the assessment of the treating physician
6. Life expectancy less than one year
7. Pregnancy or women of childbearing potential who is not sterilized or is not using a medically accepted form of contraception

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2025-01-06 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Measurement of Global longitudinal strain (GLS, %) | day 7±24 hours
  GLS adjusted for baseline.

SECONDARY OUTCOMES:
Measurement of Left ventricular ejection fraction (LVEF) | day 7±24 hours
  LVEF adjusted for baseline
Measurement of NT-proBNP (N-terminal pro b-type natriuretic peptide ) | day 7±24 hours
  NT-proBNP adjusted for baseline
Concentration of cardiac troponin-T | Day 30
  Area under the curve
Concentration of cardiac troponin-I | Day 30
  Area under the curve

OTHER OUTCOMES:
Measurement of Infarct size | Day 30
  MI size assessed by CMRI (sub-study)

CONTACTS AND LOCATIONS:
Locations (1):
- Sahlgrenska University Hospital, Gothenburg, Sweden

IPD SHARING:
Plan to Share IPD: Undecided
Plan has not be decided